CLINICAL TRIAL: NCT04525690
Title: Improving Inpatient Screening for Hepatitis C: A Stepped-Wedge Randomized Clinical Trial
Brief Title: Improving Inpatient Screening for Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 842718
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV screening; nudge; defaults
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Hospital sites will be cluster randomized to the intervention in 3 month blocks over 6 months, after which both sites will receive the default intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal study investigator and data analyst will not have knowledge of when the hospital sites are randomized to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCV Screening Default-1 Hospital Crossed Over (Experimental): Upon entering the admission order set in the EHR clinicians will receive a default order for HCV screening for eligible patients. Clinicians will have the opportunity to opt-out and not order screening
  Interventions: Behavioral: Nudge
- HCV Screening Default-2 Hospitals Crossed Over (Experimental): Upon entering the admission order set in the EHR clinicians will receive a default order for HCV screening for eligible patients. Clinicians will have the opportunity to opt-out and not order screening.
  Interventions: Behavioral: Nudge

INTERVENTIONS:
Behavioral: Nudge — Clinicians will receive a default order upon entering the the admission order set. They will have the opportunity to opt-out and not order screening. Clinicians will receive the nudge each time they enter the admission order set for a new, eligible patient.

SUMMARY:
This study will use a stepped-wedge cluster randomized clinical trial to evaluate a health system initiative to set defaults in the electronic health record admission order set to nudge inpatient hepatitis C (HCV) screening.

DETAILED DESCRIPTION:
The hepatitis C virus (HCV) is the leading cause of liver transplant and hepatocellular carcinoma in the United States, but direct-acting antiviral medications are now available and can cure the disease in over 95% of those that are treated. The Centers for Disease Control and Prevention (CDC) estimate that 75% of all chronic HCV infections in the United States are among adults born between 1945 and 1965. The CDC and US Preventive Services Task Force (USPTF) therefore recommends birth cohort screening for all adults born in this time period. In 2016, the Commonwealth of Pennsylvania signed into law a requirement that all hospitalized patients born during this time period be offered HCV screening. In this study, a stepped-wedge cluster randomized clinical trial will be conducted to test the effect of defaulting HCV screening into the admission order set to improve screening rates.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted to the Hospital of the University of Pennsylvania (HUP) or Penn Presbyterian Medical Center (PPMC)
* Born between 1945 and 1965

Exclusion Criteria:

* Patients will be excluded if they have already received Hepatitis C screening or have been previously diagnosed with Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7634 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Change in percentage of eligible patients that receive HCV antibody screening | 6 months
  The change in the percentage of eligible hospitalized patients that receive HCV antibody screening

OTHER OUTCOMES:
Percentage of patients that are HCV antibody positive | 9 months
  The percentage of eligible hospitalized patients that are HCV antibody positive
Percentage of patients that have positive HCV testing who receive either linkage to care and/or treatment | 9 months
  The percentage of eligible hospitalized patients that have positive HCV testing who receive either linkage to care and/or treatment
Change in the percentage of eligible patients that are viral load positive for HCV | 9 months
  The change in the percentage of eligible hospitalized patients that are viral load positive for HCV

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S Patel, MD, Principal Investigator — University of Pennsylvania; Shivan J Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Torgersen J, Small DS, Mallozzi CP, McGreevey JD 3rd, Rareshide CAL, Evans CN, Epps M, Stabile D, Snider CK, Patel MS. Effect of a Default Order vs an Alert in the Electronic Health Record on Hepatitis C Virus Screening Among Hospitalized Patients: A Stepped-Wedge Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e222427. doi: 10.1001/jamanetworkopen.2022.2427. PMID 35297973